CLINICAL TRIAL: NCT01568203
Title: Phase I, Randomized, Placebo-Controlled, Ascending Single Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of AMG 579 in Healthy Adult Subjects and Patients With Stable Schizophrenia or Schizoaffective Disorder
Brief Title: First-in-Human Study to Evaluate AMG 579 in Healthy Subjects and Patients With Stable Schizophrenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Amgen decision (business)
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20101275
Record Dates: First submitted 2012-02-27; First posted 2012-04-02 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Schizophrenia
Keywords: single dose, safety, healthy subjects, schizoaffective disorder, AMG 579
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — 1-(4-(3-(4-(1H-benzo(d)imidazole-2-carbonyl)phenoxy)pyrazin-2-yl)piperidin-1-yl)ethanone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 579 (Experimental)
  Interventions: Drug: AMG 579
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 579 — 3 dose levels of single oral dose administration of AMG 579 in healthy subjects (Part A), and 5 dose levels of single oral dose administration of AMG 579 in patients with schizophrenia or schizoaffective disorder (Part B)
  Arms: AMG 579
Drug: Placebo — Matching placebo control for AMG 579 at each dose level
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of AMG 579 following a single oral dose administration in healthy subjects (Part A) and in patients with schizophrenia or stable schizoaffective disorder (Part B). The study in healthy subjects (Part A) concluded, and following a protocol amendment, enrolled only patients with schizophrenia or stable schizoaffective disorder (Part B).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia (chronic, all types) or schizoaffective disorder according to Diagnostic and Statistical Manual of Mental Disorders, 4th edition Text Revision (DSM-IV-TR) criteria and by Mini International Neuropsychiatric Interview (M.I.N.I.) 6.0 for Schizophrenia and Psychotic Disorders Studies
* Body weight greater or equal to 50 kg and body mass index (BMI) between 18 and 38.0 kg/m2, inclusive, at screening
* Patient is judged by the Investigator to be likely to tolerate being off of antipsychotic medications for the duration of the trial (for patients withdrawing from or currently not taking antipsychotic medications)
* Clinically stable, as judged by the investigator, and in a non-acute phase for at least 12 weeks within enrollment. If patient is on antipsychotic medications, they must be on second generation oral antipsychotic therapy (eg, ziprasidone, quetiapine, olanzapine, etc) for at least 8 weeks within enrollment and at least one month within enrollment on a stable dose

Exclusion Criteria:

* Hospitalized for psychiatric symptoms in the 3 months within enrollment
* Patients with evidence of mental retardation by history or clinical examination or known premorbid IQ ≤ 70
* Current risk of self-harm or violence as determined by the investigator, or current risk of suicide or history of suicidal behavior within 12 months of enrollment, and/or ongoing suicidal ideation as assessed using Columbia-Suicidal Severity Rating Scale (C-SSRS) at screening (eg, any response of "yes" to the Suicidal Ideation questions on the C-SSRS in the past 12 months).

Additional critera apply. Eligibility criteria for healthy subjects (Part A) not outlined above.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Number of adverse events per subject to include clinically significant changes in neurological examinations, safety laboratory tests, electrocardiograms, and vital signs | Up to 15 days
Incidence of treatment-emergent suicidal ideation and behavior | Up to 15 days
  Measured by Columbia-Suicide Severity Rating Scale (C-SSRS)

SECONDARY OUTCOMES:
Peak plasma and cerebrospinal fluid (CSF; cohort 4 healthy subjects only) concentration (Cmax) of AMG 579 | Up to 15 days
Time of peak plasma and CSF (cohort 4 only healthy subjects only) concentration (tmax) of AMG 579 | Up to 15 days
Area under the plasma and CSF (cohort 4 healthy subjects only) concentration versus time curve (AUC) of AMG 579 | Up to 15 days
Terminal phase half-life (t1/2) in plasma and CSF (cohort 4 healthy subjects only) of AMG 579 | Up to 15 days
Scores on Simpson Angus Scale (SAS) and Barnes Akathesia Rating Scale (BARS) | Up to 15 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Glendale, California, United States

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com